CLINICAL TRIAL: NCT00509587
Title: A Phase 2 Study of GW786034 (Pazopanib) in Patients With Recurrent and/or Metastatic Invasive Breast Carcinoma
Brief Title: Pazopanib in Treating Patients With Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00199; NCI-2009-00199 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000557347; PHL-057; PHL-057 (Other: University Health Network-Princess Margaret Hospital); 7638 (Other: CTEP); N01CM62203 (NIH)
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pazopanib

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive oral pazopanib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pazopanib hydrochloride; Procedure: pharmacological study; Procedure: laboratory biomarker analysis

INTERVENTIONS:
Drug: pazopanib hydrochloride — Given orally
  Other Names: GW786034B; Votrient
Procedure: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Procedure: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving pazopanib works in treating patients with recurrent or metastatic invasive breast cancer. Pazopanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the antitumor activity of pazopanib, in terms of objective response rate (partial and complete response), in patients with recurrent or metastatic invasive breast cancer.

SECONDARY OBJECTIVES:

I. To determine the duration of objective response, rate and duration of stable disease.

II. To determine 6-month progression-free and median and overall survival rates in patients treated with this drug.

III. To document the safety and tolerability of this drug in these patients.

OUTLINE: This is a multicenter, open label study.

Patients receive oral pazopanib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Blood samples are collected at baseline and at 1, 4, and 8 weeks for correlative laboratory studies. Blood samples are evaluated for the following tumor markers by ELISA: VEGF, bFGF, sFLT-1, sTIE-2, sE-Selectin, VCAM-1, PDGF-AA, PDGF-AB and PDGF-BB. TSP-1 in plasma is measured by Accucyte™ competitive immunoassay.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Criteria:

* No prior bevacizumab
* Histologically or cytologically confirmed invasive breast carcinoma (recurrent or metastatic disease)
* Measurable disease, defined as >= 1 unidimensionally measurable lesion >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan
* Patients who may still benefit from hormonal therapy are ineligible (patients with hormone receptor-positive breast cancer should have received appropriate sequential hormonal therapy for metastatic disease until disease progression)
* Patients with HER-2 positive disease who have not yet received trastuzumab (Herceptin®) to maximal benefit are ineligible (patients with disease progression during trastuzumab therapy are eligible)
* No known brain metastases
* ECOG performance status (PS) 0-1 or Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Absolute neutrophil count >= 1,500/mm³
* Platelets >=100,000/mm³
* Total bilirubin normal (exception made for patients with known Gilbert's disease)
* AST/ALT =< 2.5 times upper limit of normal (ULN)
* No proteinuria > +1 on two consecutive dipsticks taken >= 1 week apart
* PT/INR/PTT =< 1.2 times ULN
* No allergic reactions attributed to compounds of similar chemical or biologic composition to pazopanib or other study agents
* No QTc prolongation (defined as a QTc interval >= 500 msecs) or other significant ECG abnormalities
* No condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, or active peptic ulcer disease) that would impair ability to swallow and retain study drug
* No poorly controlled hypertension (systolic blood pressure [BP] >= 140 mm Hg or diastolic BP >= 90 mm Hg) Initiation or adjustment of BP medication is allowed prior to study entry provided that the average of 3 BP readings prior to study entry is < 140/90 mm Hg
* No serious or non-healing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the last 4 weeks
* No cerebrovascular accident within the last 6 months
* No myocardial infarction, cardiac arrhythmia, hospital admission for unstable angina within the last 12 weeks
* No venous thrombosis within the last 12 weeks
* No NYHA class III-IV heart failure Patients with a history of class II heart failure may be considered eligible provided they are asymptomatic on treatment
* No concurrent uncontrolled illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C), radiotherapy, or surgery
* No cardiac angioplasty or stenting within the last 12 weeks
* No more than 1 prior chemotherapy regimen for recurrent disease
* No prior surgical procedures affecting absorption
* No CYP2C9 substrates during or for 1-2 weeks after completion of study treatment, including any of the following:

Therapeutic warfarin Low molecular weight heparin or prophylactic low-dose warfarin are allowed

* No CYP2C9 substrates during or for 1-2 weeks after completion of study treatment, including any of the following:

  * Erectile dysfunction agents: sildenafil, tadalafil, or vardenafil
  * Antiarrhythmics: bepridil, flecainide, lidocaine, mexilitine, amiodarone, or quinidine
  * Immune modulators: cyclosporine, tacrolimus, or sirolimus
  * Miscellaneous: theophylline, quetiapine, or risperidone
* No CYP2C9 substrates during or for 1-2 weeks after completion of study treatment, including any of the following:

  * Oral hypoglycemics: glipizide, glyburide, or tolbutamide
  * Ergot derivatives: dihydroergotamine, ergonovine, ergotamine, or methylergonovine
  * Neuroleptics: pimozide
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* WBC >= 3,000/mm³
* No more than 2 prior palliative systemic chemotherapy regimens for de novo metastatic disease
* Creatinine normal OR creatinine clearance >= 60 mL/min
* At least 3 months since prior trastuzumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (3):
- Canada (3):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - The Ottawa Hospital Cancer Centre (Ottawa Health Research Institute) Civic Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pazopanib Hydrochloride)
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 54 [33 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Partial and Complete Response.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT / MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 3 years
Measure: Number; unit: participant
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 21
participant | 1

2. Secondary Outcome: Duration of Objective Response
Time Frame: From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 3 years
Population: Duration of objective response was not analyzed for 1 patient who achieved PR
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Stable Disease
Time Frame: From the start of the treatment until the criteria for progression are met, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 21
months | 5.3 [2 to 20]

4. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a nontarget lesion, or the appearance of new lesions
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 21
percentage of patients | 22 [8 to 58]

5. Secondary Outcome: Overall Survival
Description: Computed using the Kaplan-Meier method.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 21
months | 12.8 [7.6 to NA] — Upper bound was not reached, as too few events

6. Secondary Outcome: Adverse Events Graded According to the NCI CTCAE Version 3.0
Description: grade 3- 4 toxicities - transaminitis, hypertension, and neutropenia in three patients each (14% each) and grade 3 gastrointestinal hemorrhage in one patient (5%).
Time Frame: Up to 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 21
percentage of patients
  Grade 3-4 transaminitis | 14
  Grade 3-4 Hypertension | 14
  Grade 3-4Neutropenia | 14
  Grade 3 gastrointestinal hemorrhage | 5

ADVERSE EVENTS:
Arm/Group | Treatment (Pazopanib Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pazopanib Hydrochloride) (N=21)
Intra abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pazopanib Hydrochloride) (N=21)
Hypertension (Vascular disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 13 (13)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Neutrophil Count decreased (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less